CLINICAL TRIAL: NCT04579146
Title: ROLE OF IMMUNE ACTIVATION PROFILES IN CORONARY ATHEROTHROMBOSIS IN PATIENTS HIV-1-INFECTED ON EFFECTIVE ANTIRETROVIRAL THERAPY
Brief Title: Coronary Artery Disease (CAD) in Patients HIV-infected
Acronym: CoroVIH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hôpital Européen Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A00219-48
Record Dates: First submitted 2020-09-24; First posted 2020-10-08 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIV-1 patients and treated effectively for more than 12 months: X-ray examination with contrast by a 64-slice CT coronary angiography.
  Interventions: Other: coronary computed tomographic angiographic (CCTA)

INTERVENTIONS:
Other: coronary computed tomographic angiographic (CCTA) — x-ray examination with contrast by a 64-slice CT coronary angiography.

SUMMARY:
HIV-infected patients with intermediate-high risk have a high prevalence of CAD and a substantial proportion of obstructive CAD. Degree of stenosis is associated with immunoactivation (lymphocyte and monocyte) and microbial translocation

ELIGIBILITY:
Inclusion Criteria:

HIV-infected patients >= 45 years with 2 or more CV risk factors currently on ART HIV-RNA < 50 copies >= 12 months (one blip allowed) Asymptomatic regarding cardiac symptoms (chest pain, syncope, dyspnea) Stable ART for more than 6 months

Exclusion Criteria:

* Sign of coronary pathology (chest pain, syncope, dyspnea).
* ATCD of allergy to IV contrast agents
* Chronic inflammatory disease other than HIV
* Subject to a measure for the protection of justice

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient VIH-1
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-09-07 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
correlation between a particular profile of immune activation in patients HIV under treatment presenting cardiovascular risk factors and the presence of coronary atheromatous plaques | 24 months
  Assessment of the prevalence of obstructive coronary artery disease in patients infected with HIV and asymptomatic with a 64-slice CT coronary angiography.

SECONDARY OUTCOMES:
Identify the bacterial populations constituting the intestinal microbiota in patients infected with HIV and look for a microbiotic signature in patients with subclinical atherothrombosis. | 24 months
  microbial translocation (16S DNA)

CONTACTS AND LOCATIONS:
Locations (1):
- BENNANI, Marseille, France

IPD SHARING:
Plan to Share IPD: No